CLINICAL TRIAL: NCT04655755
Title: A Phase I/II Study of Venetoclax in Combination With ASTX727 (Cedazuridine/Decitabine) in Treatment-Naïve High-Risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Venetoclax in Combination With ASTX727 for the Treatment of Treatment-Naive High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0129; NCI-2020-09915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0129 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ASTX727) (Experimental): Patients receive venetoclax orally PO QD on days 1-14. Patients also receive ASTX727 PO QD on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; Inqovi
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial studies the side effects and best dose of venetoclax in combination with cedazuridine and decitabine (ASTX727) in treating patients with high risk myelodysplastic syndrome or chronic myelomonocytic leukemia who have not received prior treatment (treatment-naive). Chemotherapy drugs, such as venetoclax, cedazuridine, and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability (phase 1) and overall response rate (ORR) (phase 2) of venetoclax in combination with ASTX727 in patients with treatment-naive high-risk myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) with bone marrow excess blasts > 5%.

SECONDARY OBJECTIVES:

I. Rate of complete remission (CR). II. Rate of marrow/morphologic complete remission (mCR). III. Rate of hematologic improvement (HI; erythroid/platelet/neutrophil responses).

IV. Rate of red blood cell (RBC) transfusion independence. V. Rate of platelet (PLT) transfusion independence. VI. Rate of cytogenetic response. VII. Rate of bone marrow blast response. VIII. Time to transformation to acute myeloid leukemia (AML). IX. Duration of response (DOR). X. Overall survival (OS). XI. Progression-free survival (PFS). XII. Disease-free survival (DFS). XIII. Time to next MDS treatment (TTNT). XIV. Event-free survival (EFS).

EXPLORATORY OBJECTIVE:

I. To investigate the effects of therapy on MDS and to identify biological markers of response to venetoclax and/or its combination with ASTX727.

OUTLINE: This is a phase I, dose-escalation study of venetoclax, followed by a phase II study.

Patients receive venetoclax orally (PO) once daily (QD) on days 1-14. Patients also receive ASTX727 PO QD on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment-naive high-risk (HR)-MDS or CMML (intermediate [Int]-2 or high risk by the International Prognostic Scoring System [IPSS] with overall score >= 1.5) with excess blasts > 5. Note: Patients with therapy-related MDS are eligible. Hydroxyurea is allowed to lower the white cell count =< 10,000/ul prior to initiation of venetoclax
* Total bilirubin < 3 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 3.0 x ULN unless considered due to leukemic involvement
* Creatinine < 2 x ULN unless related to the disease
* Signed written informed consent
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment
* Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment
* Age >= 18 years of age

Exclusion Criteria:

* Patients having received any prior BCL2 inhibitor therapy
* Patients with MDS with IPSS risk categories low or Int-1 (overall IPSS score < 1.5)
* Patient with known human immunodeficiency virus (HIV) infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax). HIV testing will be performed at screening, only if required per local guidelines or institutional standards
* Patient known to be positive for hepatitis B or C infection (hepatitis C virus antibody [HCV Ab] indicative of a previous or current infection; and/or positive hepatitis B surface antigen [HBs Ag] or detected sensitivity on hepatitis B virus-deoxyribonucleic acid [HBV-DNA] polymerase chain reaction [PCR] test for hepatis B core antibody [HBc Ab] and/or HBs Ab positivity) with the exception of those with an undetectable viral load within 3 months of screening. (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate
* Patient has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment
* Patient has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment
* Patient has a cardiovascular disability status of New York Heart Association class > 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain
* Patient has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition or known hypersensitivity to any of the study medications including excipients of azacitidine that in the opinion of the investigator would adversely affect his/her participating in this study
* Patient has a malabsorption syndrome or other condition that precludes enteral route of administration
* Patient exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal)
* Patient has received a live attenuated vaccine within 4 weeks prior to the first dose of study drug
* Patient has a history of other malignancies within 2 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; requires discussion with TA MD
* Patient has a white blood cell count > 25 x 10^9/L. (Hydroxyurea or leukapheresis are permitted to meet this criterion)
* Female subject has positive results for pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of all reported adverse events (Phase I) | Up to 28 days
  The overall incidence and severity of all reported adverse events using Common Toxicity Criteria version 5.0.
Overall response rate (ORR) (Phase II) | Up to 8 weeks
  ORR will be defined as the proportion of patients who had complete remission (CR), partial remission (PR) or marrow CR (mCR), or hematologic improvement (HI) lasting at least 8 weeks. Will estimate the ORR for the combination treatment, along with the 95% credible interval.

SECONDARY OUTCOMES:
Rate of complete remission | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of marrow/morphologic complete remission | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of hematologic improvement (HI; erythroid/platelet/neutrophil responses) | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of red blood cell transfusion independence | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of platelet transfusion independence | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of cytogenetic response | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Rate of bone marrow blast response | Up to 5 years post treatment
  Will be estimated with the 95% credible interval.
Duration of response | From the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first, assessed up to 5 years
Time to transformation to acute myeloid leukemia | Up to 5 years post treatment
  Time to transformation to acute myeloid leukemia is defined as the period from treatment till transformed to acute myeloid leukemia.
Overall survival | From treatment start till death, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier.
Progression-free survival | From treatment start till disease progression or death, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier.
Disease-free survival | Up to 5 years post treatment
Time to next myelodysplastic syndrome (MDS) treatment | From initial treatment start till the next MDS treatment, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier.
Event-free survival | From treatment initiation to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier.

OTHER OUTCOMES:
Biomarker analysis | Up to 5 years post treatment
  The association between cellular biomarker, and antitumor activity will be compared using Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bataller A, Montalban-Bravo G, Bazinet A, Alvarado Y, Chien K, Venugopal S, Ishizawa J, Hammond D, Swaminathan M, Sasaki K, Issa GC, Short NJ, Masarova L, Daver NG, Kadia TM, Colla S, Qiao W, Huang X, Kanagal-Shamanna R, Hendrickson S, Ravandi F, Jabbour E, Kantarjian H, Garcia-Manero G. Oral decitabine plus cedazuridine and venetoclax in patients with higher-risk myelodysplastic syndromes or chronic myelomonocytic leukaemia: a single-centre, phase 1/2 study. Lancet Haematol. 2024 Mar;11(3):e186-e195. doi: 10.1016/S2352-3026(23)00367-8. Epub 2024 Feb 2. PMID 38316133
- See also: MD Anderson Cancer Center — http://www.mdanderson.org